CLINICAL TRIAL: NCT01116557
Title: CARTO® 3 System-guided RF Ablation Using the THERMOCOOL® Catheter Versus Fluoroscopy-guided RF Ablation Using the Pulmonary Vein Ablation Catheter® (PVAC®) in Subjects With Paroxysmal Atrial Fibrillation: A Prospective, Multi-center, Randomized (2:1), Controlled, Two-arm, Unblinded Clinical Study
Brief Title: Efficacy, Safety and Efficiency Study of CARTO® 3 System Guided THERMOCOOL® Catheter Ablation Versus Fluoroscopy Guided Ablation With the Pulmonary Vein Ablation Catheter® (PVAC®)
Acronym: CLARITY-AF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Biosense stopped Study enrollment following publications that reported PVAC ablation is linked with a higher incidence of asymptomatic cerebral embolic lesions
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: BWI130
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
Keywords: radiofrequency; ablation; atrial fibrillation; CARTO; THERMOCOOL; LASSO; PVAC
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- THERMOCOOL® group (Other): Radiofrequency ablation to achieve PVI using the CARTO® 3 System, the THERMOCOOL® Catheter and the LASSO® Circular Mapping Catheter.
  Interventions: Device: Radiofrequency Ablation procedure
- PVAC® group (Active Comparator): Radiofrequency ablation to achieve PVI using fluoroscopy and the PVAC®
  Interventions: Device: Radiofrequency Ablation procedure

INTERVENTIONS:
Device: Radiofrequency Ablation procedure — Radiofrequency Ablation procedure Application of radiofrequency energy with the THERMOCOOL® catheter used in combination with the CARTO® 3 System and the LASSO® Circular Mapping Catheter to eliminate potentials arising from the pulmonary veins.
  Other Names: CARTO®3 System; LASSO® Circular Mapping Catheter; THERMOCOOL® Catheter
  Arms: THERMOCOOL® group
Device: Radiofrequency Ablation procedure — Application of radiofrequency energy with the Pulmonary Vein Ablation Catheter® (PVAC®) to eliminate potentials arising from the pulmonary veins.
  Other Names: PVAC®
  Arms: PVAC® group

SUMMARY:
The purpose of this study is to compare the efficacy, safety and efficiency of CARTO® 3 system guided THERMOCOOL® catheter ablation and fluoroscopy guided Pulmonary Vein Ablation Catheter® (PVAC®) guided ablation for the treatment of paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, randomized (2:1), controlled, two-arm, unblinded, clinical study, which will evaluate the efficacy, safety, and efficiency of CARTO® 3 System-guided RF ablation (using the THERMOCOOL® Catheter and LASSO® Circular Mapping Catheter) compared to fluoroscopy-guided RF ablation (using the PVAC®). Patients with symptomatic PAF who meet the inclusion criteria will be considered for study participation and may be enrolled if no exclusion criteria apply.

Eligible subjects who signed the study informed consent form will be randomized into one of two treatment groups:

* THERMOCOOL® Group: RF ablation to achieve PVI using the CARTO® 3 System, THERMOCOOL® Catheter and LASSO® Circular Mapping Catheter
* PVAC® Group: RF ablation to achieve PVI using fluoroscopy and the PVAC®

ELIGIBILITY:
Inclusion Criteria:

* Patients with PAF who have had two (2) symptomatic PAF episodes in the six (6) months prior to randomization, and who are selected for catheter ablation for the treatment of their AF. Additionally patients with recurrent AF with episodes up to 30 days with sinus rhythm maintained for more than one week following cardioversion and who require PVI only for the treatment of their AF (supported by the consensus statement2). At least one AF episode should be documented either on ECG, TTM, HM or telemetry strip.
* Failure of at least one AAD for PAF [class I or III] as evidenced by recurrent symptomatic PAF, or intolerable side effects due to the AAD.
* Signed Patient Informed Consent Form.
* Age 18 years or older.
* Able and willing to comply with all pre- and follow-up testing and requirements.

Exclusion Criteria:

* Longstanding persistent atrial fibrillation
* Patients with a history of any atrial flutter requiring ablation in the right atrium during the study procedure
* Patients in whom sinus rhythm was maintained for less than 1 week after electrical cardioversion
* Previous ablation for AF
* LA size > 55 mm
* LVEF < 40% (ejection fraction)
* AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause
* CABG procedure within the last six (6) months
* Awaiting cardiac transplantation or other cardiac surgery
* Documented left atrial thrombus on imaging (eg, TEE)
* Diagnosed atrial myxoma
* Women who are pregnant (by history of menstrual period or pregnancy test if the history is considered unreliable) or breastfeeding
* Acute illness or active systemic infection or sepsis
* Unstable angina
* Uncontrolled heart failure
* Myocardial infarction within the previous two (2) months
* History of blood clotting or bleeding abnormalities
* Contraindication to anticoagulation therapy (ie. heparin or warfarin)
* Life expectancy less than 12 months
* Enrollment in any other study evaluating another device or drug
* Presence of intramural thrombus, tumor or other abnormality that precludes catheter introduction or manipulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Freedom from documented AF/AT recurrences without new AADs | 1 year follow-up post-ablation
  Subjects will be considered a success for the primary efficacy endpoint if the subject is free from documented recurrences of AF or AT lasting more than 30s as measured with Transtelephonic Monitoring and Standard of Care arrhythmia monitoring during a 3-12 month follow-up period post-ablation.
Incidence of PV Stenosis (number of PVs with a reduction in diameter ≥ 50% at 6 months compared to baseline per CT or MRI) | at 6 months post-ablation
Total procedure time | at the time of the initial ablation procedure

SECONDARY OUTCOMES:
Acute procedural success | at the time of the initial ablation procedure
  Measured by the number (%) of subjects with confirmed entrance block at the end of the ablation procedure
Repeat ablation procedures for AF/AT recurrences | through 3-12 month follow-up period post-ablation
  Measured by % of subjects undergoing repeat ablation procedures for Recurring AF/AT
Freedom from documented AF/AT recurrences without AAD(s) | through 3-12 month follow-up period post-ablation
  Measured by % achieving freedom from documented AF/AT recurrences
Freedom from documented AF/AT recurrences with AAD(s) | through 3-12 month follow-up period post-ablation
  Measured by % achieving freedom from documented AF/AT recurrences
Freedom from documented AF/AT recurrences after more than one ablation procedure | through 3-12 month follow-up period post-ablation
  Measured by % achieving freedom from documented AF/AT recurrences
Freedom from documented AF recurrences without AADs | through 3-12 month follow-up period post-ablation
  Measured by % achieving freedom from documented AF/AT recurrences
Freedom from documented AF recurrences with AAD(s) | through 3-12 month follow-up period post-ablation
  Measured by % achieving freedom from documented AF/AT recurrences
Freedom from documented symptomatic AF/AT recurrences without new AAD(s) | through 3-12 month follow-up period post-ablation
  Measured by % achieving freedom from documented symptomatic AF/AT recurrences
Freedom from documented symptomatic AF/AT recurrences with AAD(s) | through 3-12 month follow-up period post-ablation
Incidence of any procedure-related and/or device-related adverse events occurring during the study | through 1 year follow-up
Incidence of any catheter-related adverse events | during 7 days follow-up post-ablation
Total Fluoroscopy exposure time | at the time of the ablation procedure
  Measured by fluoroscopy and cine-fluoroscopy time throughout procedure
Total Fluoroscopy Dose-Area Product/Source Intensifier Distance | at the time of the ablation procedure
Incidence of any phrenic nerve paralysis | through 1 year follow-up post-ablation
Incidence of any symptomatic Transient Ischemic Attack (TIA) or Cerebrovascular Accident (CVA) | through 1 year follow-up post-ablation
Number of mapping and ablation catheters used per subject | through 1 year follow-up post-ablation
Quality of Life (SF-36®) and Atrial Fibrillation Symptom Frequency and Severity Checklist assessment | Baseline, 3, 6 and 12 months
Total procedure hospital visit and ablation procedure costs | during hospitalization stay for study treatment
Total number of initial or prolonged hospitalizations and unscheduled arrhythmia-related health care provider visits (including emergency department visits) | through 1 year follow-up post-ablation

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Duytschaever, MD, Principal Investigator — A.Z. St Jan AV; Yves De Greef, MD, Principal Investigator — A.Z. Middelheim; Stuart Harris, MD, Principal Investigator — Essex Cardiothoracic Centre; Peter Steen Hansen, MD, Principal Investigator — Heart Center Varde; Pepijn Van Der Voort, MD, Principal Investigator — Catharina Ziekenhuis; Thomas Deneke, MD, Principal Investigator — Krankenhaus Porz Cologne; Atul Verma, MD, Principal Investigator — Southlake Regional Health Centre; Arif Elvan, MD, Principal Investigator — Isala; Yaariv Khaykin, MD, Principal Investigator — Southlake Regional Health Centre